CLINICAL TRIAL: NCT07256821
Title: A Prospective, Mixed Methods, Observational Study to Define a Diaphragm-focussed and Patient-acceptable Inspiratory Muscle Training (IMT) Load in Difficult to Wean, Mechanically Ventilated Patients
Brief Title: Identifying the Optimal IMT Dose in ICU
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25/WA/0242
Record Dates: First submitted 2025-11-18; First posted 2025-12-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Difficult to Wean, Mechanically Ventilated Patients With a Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training at no load, and at 15, 25, 35 and 45% participants maximal inspiratory pressure

SUMMARY:
200,000 adults are admitted to intensive care in the UK each year. Many of these patients need help with their breathing and are put on a machine called a ventilator.

Research shows that many patients using a ventilator quickly develop weakness in their main breathing muscle, called the diaphragm. This weakness can cause a longer time on the ventilator, a longer hospital stay, and higher chances of health problems or death.

Inspiratory muscle training is a breathing exercise where the patient breathes against resistance through a small device (like breathing through a straw). It aims to improve the strength of the diaphragm and reduce how long patients are on the ventilator.

Why is this research needed?

Research shows that current breathing exercise programmes do not help patients come off the ventilator or go home quicker. This may be because these breathing exercises strengthen the wrong muscles (those in the chest and neck, that are not efficient). These exercises can also be distressing for patients.

What will be done in this research? This research aims to develop a breathing exercise programme that focusses on strengthening the diaphragm. We will also make sure patients do not find the breathing exercise too distressing.

This research will measure how the breathing muscles respond to four different levels of breathing exercise and ask patients to feedback on each level.

1. At each breathing exercise level, the effort of the breathing muscles will be measured using a small tube inserted into the nostril and small sticky patches on the chest and neck. We aim to find the level where the diaphragm is being pushed to work hard but other muscles in the chest and neck are not.
2. After each breathing exercise level patients will be asked how they found it - for example, easy, pleasant, scary.

This procedure will be repeated 1-3 times over seven days with at least 24 hours between each measurement

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients with a tracheostomy
* Aged ≥ 18 years
* Co-operative and able to participate in IMT.
* Informed consent or surrogate approval

Exclusion Criteria:

* Facial or skull fracture, or a bleeding disorder which would prohibit oesophageal catheter placement.
* Undrained pneumothorax/pneumomediastinum.
* Delirium or deep sedation that impedes the patient's ability to participate in study procedures
* Pregnancy
* Unlikely to survive, or consultant assessment that the patient is not appropriate.
* Wounds that prohibit EMG electrode placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Difficult to wean, mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic muscle activation (measured by electromyography) | Up to 7 days
  At rest and at each IMT load on each study occasion
Extra diaphragmatic muscle activity (surface electromyography of scalene, sternocleidomastoid and parasternal muscles) | Up to 7 days
  At rest and at each IMT load on each study occasion
Perceived difficultly and unpleasantness (number rating scale 0-10) | Up to 7 days
  At each IMT load on each study occasion
The experience of IMT using qualitative techniques including verbal and non-verbal (including written communication, picture and word boards) | Up to 7 days
  At each IMT load on each study occasion

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield Hospitals, Marlow, United Kingdom

IPD SHARING:
Plan to Share IPD: No